CLINICAL TRIAL: NCT00539500
Title: Autologous Stem Cell Rescue With CD133+ Selected Hematopoietic Progenitor Cells in Patients With High-Risk Neuroblastoma
Brief Title: Autologous Stem Cell Rescue With CD133+ Selected Cells in High-Risk Neuroblastoma
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow Accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0374
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; ClinicMACS; CliniMACS; Stem Cell Transplantation; Blood And Marrow Transplantation; Pediatric; Solid Tumors; Carboplatin; Paraplatin; Etoposide; VePesid; Melphalan; Alkeran; CD133+ Cells
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Etoposide; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transplantation CD133+ cells (Experimental): Stem Cell Transplantation of CD133+ cells using the ClinicMACS in combination with Carboplatin + Etoposide + Melphalan
  Interventions: Drug: Carboplatin; Drug: Etoposide; Drug: Melphalan; Procedure: Stem Cell Infusion; Device: ClinicMACS

INTERVENTIONS:
Drug: Carboplatin — Carboplatin by vein over 24 hours for 4 days, dosing as determined at day 1.
  Other Names: Paraplatin®
Drug: Etoposide — 300 mg/m^2 by vein over 24 hours for 4 days
  Other Names: VePesid®
Drug: Melphalan — 70 mg/m^2 Intravenous Bolus for 3 Days
  Other Names: Alkeran
Procedure: Stem Cell Infusion — Stem Cell Infusion (approximately 5x10^8 TNC cells/kg CD133+ selected) on Day 0.
Device: ClinicMACS — Device used to process the blood and separate the CD 133+ cells needed for transplantation

SUMMARY:
The goal of this clinical research study is to learn how long it takes for certain types of transplanted stem cells to produce new blood cells. The safety of this treatment will also be studied. Finally, researchers want to learn if collecting the cells with the CliniMACS device can decrease the possibility of tumor cells contaminating (appearing in) the stem cells that are reinfused into participants.

DETAILED DESCRIPTION:
Researchers want to learn if a CD133+ selected autologous stem cell transplant can help to control the disease in patients with high-risk neuroblastoma. After your cells are collected, they will be treated in the cell processing lab using the CliniMACS device. This device will separate out the CD133+ cells. These selected cells will then be given back to you on the day of transplant.

If you are found to be eligible to take part in this study, you will have a small plastic tube placed in the collar bone area or the femoral vein (groin area). This is called a central venous catheter (CVC). You will sign a separate consent form for the CVC placement and the general anesthesia that is given. There may be several weeks between the collection of stem cells and the reinfusion of these cells after high-dose chemotherapy. If the CVC is placed in the femoral vein, the CVC will be removed after the stem cells are collected and a new CVC will be placed in the collar bone before you are admitted for the stem cell transplant. The CVC will be used for chemotherapy, fluids, blood products, stem cells, and other medications. The CVC will remain until it is no longer needed (usually 2-3 months).

To help move the needed stem cells from your bone marrow to your blood, a drug called granulocyte colony-stimulating factor G-CSF (filgrastim) will be injected under the skin. These injections may be given once a day for Days 2-7. You or your caregiver will be taught how to give the injections at home. After 2 days of filgrastim injections, a blood sample (about 4 teaspoons each time) will be drawn each day until you begin leukapheresis. This blood test is used to check the number of stem cells and to watch for possible side effects. You will then be instructed to either continue with the daily injections or stop. When the number of stem cells in the blood is high enough, you will go to the MD Anderson Apheresis Unit to have your stem cells collected.

The procedure to collect your stem cells is called leukapheresis. It is similar to donating platelets to a blood bank. For this procedure, the stem cells will be removed from the blood through the CVC, and the remaining blood will be given back to you through the CVC. You will have one leukapheresis procedure per day, for 1-5 days in a row, until enough stem cells are collected for the transplant. "Back-up" cells (extra cells collected during the leukapheresis procedure) will also be collected. These cells will be stored in the cell processing lab and may given back to you later if your white cell count does not recover. Each leukapheresis procedure takes about 4-6 hours. This research study will use the CliniMACS device to process the blood and separate the cells needed for transplantation. Researchers will test a small sample of the collected cells to see if any tumor cells that might be present in the blood before using the CliniMACS device are no longer present in the processed blood after using the device.

Carboplatin and etoposide are designed to interfere with the growth of cancer cells by stopping cell division, and melphalan is designed to damage the DNA (the genetic material) of cells. The combination of carboplatin, etoposide, and melphalan causes a large amount of bone marrow cells to die, which stops blood cells from being produced as normal. In order to try to restart the production of blood cells, an autologous stem cell transplant is often performed. For an autologous transplant, stem cells are removed from the blood. Usually when stem cells are collected, they are either given back to the patient as collected, or else a smaller group of cells that have a certain "marker" on their cell surface is selected (separated out) before being given back to the patient. The CliniMACS device is a machine that processes blood and separates the cells needed for transplantation. The CliniMACS device is designed to select stem cells with a different marker on the cell surface than is normally selected. The marker is called CD133+, and researchers believe that transplanting cells that have this marker will make the infused cells less likely to be contaminated with neuroblastoma cells, compared to the standard method of cell selection.

After 5 days of leukapheresis procedures, if the number of stem cells collected is lower than a certain level, you will no longer be eligible to take part in the study.

Before you can start treatment on this study, you will have "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. If these tests have been performed recently, they may not need to be repeated. To check the status of the disease, you will have CT scans, bone marrow aspirations and biopsies, and a chest x-ray. The CT scans will be performed on the chest, abdomen, and pelvis (and if needed, the brain). To collect a bone marrow biopsy, an area of the hip or chest bone is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle. You will have a pulmonary function test (to measure lung function), an echocardiogram (to measure heart function), and an electrocardiogram (EKG -- a test to measure the electrical activity of the heart). You will have a physical exam, including measurement of vital signs (such as blood pressure and heart rate), height, and weight. Blood (about 4 tablespoons) will be drawn for routine tests and to check for diseases such as hepatitis and HIV. Females who are able to have children must have a negative urine pregnancy test. You will also have a 12 or 24-hour urine test before carboplatin can be given. For this test, you will collect your urine over 12 or 24 hours. You will be provided with a container to collect the urine in. This test will be used to help decide the dosing of carboplatin that you receive.

After enough stem cells are collected, and at a time decided upon by your neuro-oncologist and transplantation doctors, you will be admitted to the hospital to receive fluids and then the chemotherapy drugs carboplatin, etoposide, and melphalan, according to the standard schedule. After the chemotherapy, you will have 3 "rest" days where no chemotherapy is given.

On the day after the third rest day, your stem cells will be infused back into your CVC. To help speed up the recovery of your white blood cells, a drug called filgrastim will be injected under the skin. You will receive a filgrastim injection under the skin once a day, until the white blood cell count recovers (usually 2-3 weeks). You may also receive standard antibiotics, fluids, and/or other medications, if your doctor feels it is necessary based on symptoms you may have. While you are in the hospital, you will have physical exams once a day. Blood (about 4 teaspoons each time) will be drawn about 3-7 days per week, until your blood counts are fully recovered and any side effects of the chemotherapy have resolved. At that time, you will be able to leave the hospital.

From the time you leave the hospital until about Day 60, you will have follow-up visits at least once per week. At these visits, you will have a physical exam. Blood (about 4 teaspoons each time) will be drawn for routine tests. However, your participation in this study will not be over until after your annual follow-up at which time you will have a medical history and physical exam, blood (about 4 teaspoons) drawn for routine tests, and a CT scan.

If the disease gets worse or intolerable side effects occur at any time in this study, you will be taken off study.

This is an investigational study. All of the drugs used in this study are commercially available and FDA approved for use in neuroblastoma. The CliniMACS device is not commercially available or FDA approved. It has been authorized for use in research only.

Up to 20 patients will take part in this study. All will be enrolled at The University of Texas (UT) MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed high-risk Neuroblastoma defined as: a. INSS 2A/2B older then 365 days with MYCN amplified, unfavorable histology, and any ploidy. b. INSS Stage 3, older than 365 days with MYCN amplification and/or unfavorable histology. c. INSS Stage 4 or 4S, less than 365 days of age, with MYCN amplification d. INSS Stage 4, over 365, regardless of MYCN amplification or histology.
2. Pre-transplant modalities may include surgery, chemotherapy, or radiation therapy. Radiation must not include lung fields. Only patients in complete response (CR), or partial response (PR) at the primary site will be eligible.
3. Any recurrent neuroblastoma with at least a partial response to salvage therapy.
4. Lansky performance score greater than or equal to 50 for patients </= 16 years of age, or Zubrod performance status score of 0-2 for patients > 16 years of age.
5. No symptomatic pulmonary disease. forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and Carbon Monoxide Diffusing Capacity (DLCO) >/= 50% of expected corrected for hemoglobin. If unable to perform pulmonary function test (most children < 6 years of age), pulse oximetry >/= 92% on room air.
6. Adequate cardiac function as demonstrated by left ventricular ejection fraction >/= 50% by echocardiogram.
7. Adequate hepatic function as defined as serum glutamic-oxaloacetic transaminase, SGOT (AST) and serum glutamic-pyruvic transaminase, SGPT (ALT)< 5 times upper limits of normal.
8. All patients and/or their parents or legal guardians must sign a written informed consent.
9. Females of childbearing potential defined as not post-menopausal for 12 months or no previous surgical sterilization must have a negative urine pregnancy test within 30 days of registering. Patients will be informed of the risk of not using adequate contraception.

Exclusion Criteria:

1. Patient is pregnant or breast-feeding.
2. Active infection not controlled by antibiotics after seven days of therapy.
3. Brain metastases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-10; Primary Completion 2012-09-05 (Actual); Study Completion 2012-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura L. Worth, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated in October of 2007 and, due to slow accrual, was closed in December 2010. All recruitment done at UT MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | Transplantation CD133+ Cells
Started | 3
Completed | 0
Not Completed | 3
Not completed — Disease Progression | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: A final summary or analysis was not possible as only 3 out of 20 planned participants were registered.
Arm/Group | Transplantation CD133+ Cells
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 4 [3 to 5]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Engraftment Failure Rate
Description: Engraftment Failure Rate is number of participants with engraftment failure out of total participants. Engraftment failure is defined as failure to achieve an absolute neutrophil count (ANC) >500/ul by day 42, and has no evidence of donor chimerism on bone marrow examination.
Time Frame: Participant evaluation at Day 42, total study up to 3 Years
Population: Study analysis not possible due to small number of participants. Of the 3 participants enrolled, 0 had engraftment failure.
Measure: Number; unit: Participant
Arm/Group | Transplantation CD133+ Cells
Number analyzed (Participants) | 3
Participant | 0

2. Secondary Outcome: Number of Participants With Device-related Toxicity Associated With Transplantation of CD133+ Cells
Description: Toxicity associated with CliniMACS device associated with transplantation of CD133+ cells in high-risk neuroblastoma. Adverse events assessed and graded according to NCI's Common Terminology Criteria for Adverse Events (CTCAE) v3.0.
Time Frame: 3 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Transplantation CD133+ Cells
Number analyzed (Participants) | 3
Participants | 3

3. Other Pre Specified Outcome: Number of Treated Participants With Engraftment Failure at Day 42
Description: Engraftment failure is defined as if by day +42 participant does not have an absolute neutrophil count (ANC) >500/ul, and has no evidence of donor chimerism on bone marrow examination.
Time Frame: Participant evaluation at Day 42
Population: Three subjects engrafted after receiving the investigational product, no other analysis available. Of the 3 participants enrolled, 0 had engraftment failure.
Measure: Number; unit: participants
Arm/Group | Transplantation CD133+ Cells
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events collected from Day -8 to Stem Cell Infusion (Day 0) through approximately Day 60 post infusion. Overall study period October 2007 to March 2011.
Arm/Group | Transplantation CD133+ Cells
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transplantation CD133+ Cells (N=3)
Anorexia (Metabolism and nutrition disorders) | 2
Nausea (Gastrointestinal disorders) | 3 (3)
Pain (Abdomen NOS) (General disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1
Distention/Bloating (Gastrointestinal disorders) | 1
Mucocitis (Clinical Exam) (Gastrointestinal disorders) | 3 (3)
Pain (Other) (General disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Febrile Neutropenia (Infections and infestations) | 1
Diarrhea (Gastrointestinal disorders) | 3 (3)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
ALT/AST Disorder (Metabolism and nutrition disorders) | 2 — aspartate transaminase (AST), alanine transaminase (ALT)
BICARBONATE, SERUM-LOW (Metabolism and nutrition disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Hemorrhage, GI (stoma) (Gastrointestinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Neuropathy: Sensory (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Bloating (Gastrointestinal disorders) | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed, rare patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No